CLINICAL TRIAL: NCT05442736
Title: Modified Surface of PLGA Nanoparticles in Smart Hydrogel: A Randomized Clinical Trial to Establish an Advanced Strategy Against Antibiotic Resistant Infections in Endodontics
Brief Title: Modified Surface of PLGA Nanoparticles in Smart Hydrogel
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Mona Gamal Mohamed Afifi Arafa, Associate Professor, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI (1643)
Record Dates: First submitted 2022-06-27; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Antibiotic Resistant Infection
Keywords: nanoparticles; endodontics infection
MeSH Terms: interventions — Ciprofloxacin; Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: Fifty-five patients having single rooted teeth with signs and/or symptoms of post treatment disease that were indicated for non-surgical root canal retreatment were participated in this study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free drug (Active Comparator): Free drug incorporated in in situ gels
  Interventions: Drug: Ciprofloxacin
- drug entrapped in nanoparticles (Active Comparator): drug entrapped in nanoparticles then incorporated in in situ gels
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — studying the effect of nanoparticles in controlling the release of the drug in addition to in situ gel
  Other Names: device

SUMMARY:
Nanoparticles containing antibiotic were prepared and incorporated in in situ gel to treat recurrent endodontic infections

DETAILED DESCRIPTION:
Enterococcus faecalis is the main cause of endodontic infections and form biofilm on dentin, resulting in treatment-resistant periradicular lesions. To overcome these problems, antibacterial nanoparticles were used because of their small size, sustained release and positive charge which interact with the negatively charged surface of bacterial cell causing its destruction. In this light, Ciprofloxacin hydrochloride (CIP) in chitosan coated PLGA nanoparticles (CIP-CS-PLGA-NPs) and free CIP were embedded in Pluronic® 407/188 to form thermosensitive gels(F1) and (F2) respectively, that were investigated in terms of viscosity, gelation temperature and in-vitro release. The antibacterial efficacy of F1 and F2 were clinically investigated on patients then compared to CIP and Ca(OH)2 pastes by determining bacterial reduction percent and biofilm inhibition assay

ELIGIBILITY:
Inclusion Criteria:

* Root canal filled single rooted teeth with post treatment disease manifested by one or more of the following signs and symptoms:
* History of recurrent acute and/or chronic periapical abscess
* Pain on palpation and/or percussion at least after one month of previous procedure
* Radiographic evidence of bone loss either as a new developing lesion or an increase in the size of a pre-existing one.

Exclusion Criteria:

* Teeth that were badly broken down indicated for extraction or with difficult isolation
* Immuno-compromised patients.
* Patients with history of taking antibiotics orally.
* Periodontally affected teeth.

Ages: 40 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2022-04-02 (Actual); Primary Completion 2022-04-16 (Actual); Study Completion 2022-04-16 (Actual)

PRIMARY OUTCOMES:
controlled release of the drug with associated with infection inhibition | two weeks
  drug entrapped in nanoparticles incorporated in in situ gel inhibited the biofilm formation and bacterial recurrent infection

CONTACTS AND LOCATIONS:
Overall Officials: Mona Arafa, Principal Investigator — The British University in Egypt
Locations (1):
- Mona Arafa, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fereig SA, El-Zaafarany GM, Arafa MG, Abdel-Mottaleb MMA. Tackling the various classes of nano-therapeutics employed in topical therapy of psoriasis. Drug Deliv. 2020 Dec;27(1):662-680. doi: 10.1080/10717544.2020.1754527. PMID 32393082